CLINICAL TRIAL: NCT02867189
Title: Developing an Atlas to Teach Nurses to Clean Micro-instruments Used in Cataract
Brief Title: Developing an Atlas to Teach Nurses to Clean Micro-instruments Used in Cataract Surgery: Effect on Patient Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hua Liu (Other)
Responsible Party: Sponsor-Investigator, Hua Liu, charge of nursing department, Tianjin Medical University Eye Hospital
Organization: Tianjin Medical University Eye Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: tjykdxykyy5
Record Dates: First submitted 2016-08-02; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2015-10

CONDITIONS: Cataract
Keywords: anterior chamber flare; cataract; intraocular pressure; micro-instrument; photograph-based atlas; visual; training nurse
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- atlas of micro-instrument (Experimental): anterior chamber cell counts and visual and intraocular pressures on postoperative days 1,3,7,14 by atlas of micro-instrument training method.
  Interventions: Other: atlas of micro-instrument
- traditional training (No Intervention): anterior chamber cell counts and visual and intraocular pressures on postoperative days1,3,7,14 by traditional training method.

INTERVENTIONS:
Other: atlas of micro-instrument — Nurses after training can improve the instrument cleaning quality, reduce the reaction after cataract surgery
  Arms: atlas of micro-instrument

SUMMARY:
Aims and objectives The purpose of this study was to develop an atlas to explore the effect of micro-instrument cleaning on the safety of cataract surgery.

Background Cataract surgery safety is affected by many factors, the most influential of which is the quality of instrument cleaning. Previous studies focused on the reaction in the eye after cataract surgery. None offered a solution for manually cleaning ophthalmic micro-instruments or response data for surgical instruments after cataract surgery.

Design The study was designed to collect quantitative data derived from postoperative ocular evaluation.

Methods We developed an atlas that details micro-instrument cleaning that could be used to train nurses to have this skill. A total of 120 cataract patients were divided evenly into experimental and control groups. In the experimental group, cataract surgery was undertaken using microsurgical instruments that were cleaned by the atlas-trained nurses. In the control group, micro-instruments were used that had been cleaned by non-atlas-trained nurses. All the patients underwent the same postoperative tests: anterior chamber cell counts and visual and intraocular pressures on postoperative days (PODs) 1, 3, 7, and 14.

DETAILED DESCRIPTION:
A single surgeon conducted all of the surgery and follow-up all patients

ELIGIBILITY:
Inclusion Criteria:

* Cataract patients

Exclusion Criteria:

* Patients with metabolic disease, immune disease, and/or retinopathy were not included in this study.

Ages: 60 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-09; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
the numbers of anterior chamber cells after cataract surgery. | within the 14 days after surgery
  the numbers of anterior chamber cell counts within the 14 days after surgery

SECONDARY OUTCOMES:
the change of vision after cataract surgery | within the 14 days after surgery
  the change of vision after cataract surgery within the 14 days after surgery

OTHER OUTCOMES:
the change of intraocular pressure after cataract surgery | within the 14 days after surgery
  the change of intraocular pressure after cataract surgery within the 14 days after surgery

IPD SHARING:
Plan to Share IPD: No